CLINICAL TRIAL: NCT05222568
Title: Effect of the Minimum Bronchial Cuff Volume of Left-sided Double-lumen Endotracheal Tube for One-lung Ventilation on the Change of the Bronchial Cuff Pressure During Lateral Positioning in Thoracic Surgery: a Prospective Observational Study
Brief Title: Effect of the Minimum Bronchial Cuff Volume of Left-sided Double-lumen Endotracheal Tube for One-lung Ventilation on the Change of the Bronchial Cuff Pressure During Lateral Positioning in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Sung Hye Byun, Assistant professor, Kyungpook National University Chilgok Hospital
Other Study IDs: KNUCH 2021-08-059-001
Record Dates: First submitted 2021-12-29; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer; Pneumothorax
Keywords: Cuff pressure; Double lumen endotracheal tube; Lateral positioning
MeSH Terms: conditions — Lung Neoplasms; Pneumothorax

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BCVmin=0: This study was a prospective observational study, and the patients was divided into two groups with BCVmin=0 or BCVmin >0, according to the BCVmin which was naturally determined during anesthesia in each patient.
  Interventions: Behavioral: Lateral positioning; Device: Cuff pressure measurement
- BCVmin>0: The patients was divided into two groups with BCVmin=0 or BCVmin >0, according to the BCVmin which was naturally determined during anesthesia in each patient.
  Interventions: Behavioral: Lateral positioning; Device: Cuff pressure measurement

INTERVENTIONS:
Behavioral: Lateral positioning — After the DLT intubation, the patient is placed in lateral decubitus position
Device: Cuff pressure measurement — The pressure of the bronchial cuff should be measured with cuff-manometer in supine position, and then measurement should be repeated after lateral positioning

SUMMARY:
Over-inflation of the bronchial cuff of the double-lumen tube (DLT) can cause damage to the airway mucosa and misplacement of the tube, and under-inflation may cause incomplete collapse of the non-ventilated lung and incomplete ventilation of the lung that should be ventilated. Appropriate cuff pressure is generally known to be ranged 20-30 cmH₂O, but in the study of Okubo et al., who observed the minimum bronchial cuff volume and pressure that did not cause air leakage using the method of confirming by capnography, it was possible to obtain the result that OLV was possible without air leakage even at a pressure lower than 25 cmH₂O (the generally recommended tube cuff pressure) in both men and women. In a recent study of Yamada et al., when using the capnography waveform-guided method to inflate the bronchial cuff by checking for air leakage using the capnography waveform, the bronchial cuff volume (BCV) that satisfies the air-tight seal was significantly smaller compared with a pressure-guided method to inflate the bronchial cuff with 20 cmH₂O.

The minimum bronchial cuff volume (BCVmin) at which such air leakage does not occur may vary from individual to individual. It is presumed that this is because the diameter of the left main bronchus (LMB) differs from individual to individual, which causes the variation of the gap between the diameter of the LMB and the outer diameter of the DLT mounted thereon. Moreover, the previous study revealed that the lateral positioning could increase the pressure of the bronchial cuff mounted on the LMB due to the gravity-induced morphological and conformational change of the trachea. Considering these factors, the researchers hypothesized that the change in the bronchial cuff pressure (BCP) due to a positional change might vary depending on whether the bronchial cuff was inflated, that is, the initially established BCVmin.

Therefore, in this study, the researchers tried to investigate the effect of BCVmin on the change of minimum bronchial cuff pressure (BCPmin) due to the positional change from the supine to lateral decubitus, by dividing the groups whose BCVmin is 0 ml or exceeds 0 ml.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-80 and with an American Society of Anesthesiologists (ASA) physical status of 1 or 3 who are scheduled to undergo elective video-assisted thoracoscopic surgery (VATS)

Exclusion Criteria:

A. Need for a right-sided DLT B. An intraluminal lesion in the left main bronchus C. An anatomical problem in the tracheobronchial tree D. Patients with chronic obstructive pulmonary disease with impaired lung compliance E. Patients with interstitial lung disease with severe pulmonary dysfunction F. Patients with Body mass index (BMI) ≥ 30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The researcher contacts patients who are potential candidates for the study at the time of their preoperative visit. The participants are being enrolled in the study at the tertiary university hospital in Daegu, South Korea, from October 2021 to December 2021
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The change in minimum bronchial cuff pressure (BCPmin) when changing a posture from supine to lateral decubitus, that is the diffence in BCPmin between the supine and lateral position when injecting the BCVmin of air. | 1. In supine position, 2 minutes after the completion of confirming the double-lumen endotrachial tube (DLT) position via fiberoptic bronchoscope (FOB), 2. In lateral position, 2 minutes after the completion of confirming the DLT position via FOB
  The bronchial cuff pressure measured when the bronchial cuff was inflated with the smallest bronchial cuff volume without air leakage was defined as BCPmin. It should be measured at each position (supine and lateral decubitus position). To do this, the bronchial cuff should be inflated with air, increasing the volume by 0.5 ml from 0 ml, and at the same time check and measure whether air is leaking around the bronchial cuff. As a method of checking for air leakage, the investigators should check whether 80% or more of the tidal volume set on the ventilator at each stage is properly supplied to the patient while increasing the air by 0.5 ml, and whether the end-tidal carbon dioxide graph has a typical trapezoidal shape.

SECONDARY OUTCOMES:
The minimum bronchial cuff volume (BCVmin) | 1. In supine position, 2 minutes after the completion of confirming the DLT position via FOB, 2. In lateral position, 2 minutes after the completion of confirming the DLT position via FOB
  The smallest bronchial cuff volume without air leak was defined as BCVmin. It should be measured at each position (supine and lateral decubitus positon). To do this, the bronchial cuff should be inflated with air, increasing the volume by 0.5 ml from 0 ml, and at the same time check and measure whether air is leaking around the bronchial cuff. As a method of checking for air leakage, the investigators should check whether 80% or more of the tidal volume set on the ventilator at each stage is properly supplied to the patient while increasing the air by 0.5 ml, and whether the end-tidal carbon dioxide graph has a typical trapezoidal shape.
The relationship between the minimum bronchial cuff volume (BCVmin) and the gap between the diameter of patient's left main bronchus and the outer diameter of the DLT | In supine position, , 2 minutes after the completion of confirming the DLT position via FOB
The incidence of the patients whose BCPmin when changing posture from supine to lateral decubitus | 1. In supine position, 2 minutes after the completion of confirming the DLT position via FOB, 2. In lateral position, 2 minutes after the completion of confirming the DLT position via FOB
  Increase or decrease of the BCPmin after positional change

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hye Byun, M.D., Principal Investigator — Kyungpook National University Chilgok Hospital
Locations (1):
- Sung Hye Byun, Daegu, South Korea

REFERENCES:
- [Background] Tobias JD. Pediatric airway anatomy may not be what we thought: implications for clinical practice and the use of cuffed endotracheal tubes. Paediatr Anaesth. 2015 Jan;25(1):9-19. doi: 10.1111/pan.12528. Epub 2014 Sep 20. PMID 25243638
- [Background] Kim JH, Kim E, Kim IY, Choi EJ, Byun SH. Changes in the Bronchial Cuff Pressure of Left-Sided Double-Lumen Endotracheal Tube by Lateral Positioning: A Prospective Observational Study. J Clin Med. 2021 Apr 9;10(8):1590. doi: 10.3390/jcm10081590. PMID 33918748
- [Background] Yuceyar L, Kaynak K, Canturk E, Aykac B. Bronchial rupture with a left-sided polyvinylchloride double-lumen tube. Acta Anaesthesiol Scand. 2003 May;47(5):622-5. doi: 10.1034/j.1399-6576.2003.00102.x. PMID 12699525
- [Background] Hannallah MS, Benumof JL, McCarthy PO, Liang M. Comparison of three techniques to inflate the bronchial cuff of left polyvinylchloride double-lumen tubes. Anesth Analg. 1993 Nov;77(5):990-4. doi: 10.1213/00000539-199311000-00020. PMID 8214739
- [Background] Sultan P, Carvalho B, Rose BO, Cregg R. Endotracheal tube cuff pressure monitoring: a review of the evidence. J Perioper Pract. 2011 Nov;21(11):379-86. doi: 10.1177/175045891102101103. PMID 22165491
- [Background] Okubo H, Kawasaki T, Shibayama A, Sata T. [Measurement of the Minimum Pressure in the Bronchial Cuff during One-lung Ventilation Using a Capnometer]. Masui. 2015 Aug;64(8):794-8. Japanese. PMID 26442408
- [Background] Yamada Y, Tanabe K, Nagase K, Ishihara T, Iida H. A Comparison of the Required Bronchial Cuff Volume Obtained by 2 Cuff Inflation Methods, Capnogram Waveform-Guided Versus Pressure-Guided: A Prospective Randomized Controlled Study. Anesth Analg. 2021 Mar 1;132(3):827-835. doi: 10.1213/ANE.0000000000005179. PMID 33002924